CLINICAL TRIAL: NCT06137989
Title: Two-year Clinical Performance of Dual- and Light-cure Bulk-fill Resin Composites in Class ӀӀ Restorations: A Randomized Clinical Trial
Brief Title: Clinical Performance of Dual- and Light-cure Bulk-fill Resin Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elshirbeny Mohamed Elawsya, Lecturer, Department of Conservative Dentistry, Faculty of Dentistry, Mansoura University, Mansoura, Egypt, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01150620
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries Class II
Keywords: Bulk-fill resin composite; Dual-cure; Light-cure; Class ӀӀ restorations; Clinical performance; Randomized clinical trial

STUDY DESIGN:
Intervention Model Description: Each patient received three Class ӀӀ restorations with the three tested bulk-fill resin composites.
Who Masked: Participant, Outcomes Assessor
Masking Description: Except the investigator, the participants and the two clinical examiners were blinded to the type of bulk-fill resin composite applied in each tooth (a double-blinded clinical trial).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fill-Up (Active Comparator): Bulk-fill resin composite type
  Interventions: Procedure: Fill-Up Class ӀӀ restoration
- QuiXfil (Active Comparator): Bulk-fill resin composite type
  Interventions: Procedure: QuiXfil Class ӀӀ restoration
- Tetric N-Ceram Bulk Fill (Active Comparator): Bulk-fill resin composite type
  Interventions: Procedure: Tetric N-Ceram Bulk Fill Class ӀӀ restoration

INTERVENTIONS:
Procedure: Fill-Up Class ӀӀ restoration — Bulk-fill technique
  Arms: Fill-Up
Procedure: QuiXfil Class ӀӀ restoration — Bulk-fill technique
  Arms: QuiXfil
Procedure: Tetric N-Ceram Bulk Fill Class ӀӀ restoration — Bulk-fill technique
  Arms: Tetric N-Ceram Bulk Fill

SUMMARY:
This study (a double-blinded, prospective, randomized clinical trial) aimed to evaluate 2-year clinical performance of dual- and light-cure bulk-fill resin composites in Class ӀӀ restorations.

The null hypothesis tested in this study was that, there would be no difference in the 2-year clinical performance of all tested bulk-fill resin composites in Class II restorations.

Forty patients were enrolled in the study. Each patient received three bulk-fill resin composites Class ӀӀ restorations. One dual-cure and two light-cure bulk-fill resin composites were used for Class ӀӀ restorations following manufacturer's instructions. A universal adhesive was used with all restorations. All restorations were clinically evaluated after 1 week (baseline), 6 months, 12 months, 18 months and finally after 24 months using the FDI World Dental Federation criteria.

ELIGIBILITY:
Inclusion Criteria:

* each participant should have at least three permanent molars and premolars that need to be treated with Class II restorations due to primary carious lesions.
* all participants required to have a full and normal occlusion and to maintain adequate oral hygiene.

Exclusion Criteria:

General exclusion criteria:

* heavy bruxism.
* poor oral hygiene.
* chronic or severe periodontitis.
* a history of allergies to any of the materials utilized in this study.
* pregnant or nursing females.

Specific exclusion criteria:

* fractured or visibly cracked teeth.
* rampant caries.
* faulty restoration opposite or adjacent to the tooth to be restored.
* atypical extrinsic staining.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Esthetic properties (FDI criteria) | From baseline to 2-year follow-up
  Including five parameters (surface luster, margin staining, surface staining, color match & translucency, and esthetic anatomical form).
  Each parameter is exhibited by five scores (1, 2, 3, 4, 5), score 1 is the best outcome.
  Three scores for acceptable (1, 2, 3) and two scores for non-acceptable (4 for reparable and 5 for replacement).
Functional properties (FDI criteria) | From baseline to 2-year follow-up
  Including five parameters (marginal adaptation, occlusal wear, proximal contact, radiographic examination, and fracture of material & retention).
  Each parameter is exhibited by five scores (1, 2, 3, 4, 5), score 1 is the best outcome.
  Three scores for acceptable (1, 2, 3) and two scores for non-acceptable (4 for reparable and 5 for replacement).
Biological properties (FDI criteria) | From baseline to 2-year follow-up
  Including three parameters (post-operative sensitivity, recurrence of caries, and tooth integrity).
  Each parameter is exhibited by five scores (1, 2, 3, 4, 5), score 1 is the best outcome.
  Three scores for acceptable (1, 2, 3) and two scores for non-acceptable (4 for reparable and 5 for replacement).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Mansoura, Egypt., Al Mansurah, Aldakhlia, Egypt